CLINICAL TRIAL: NCT02549482
Title: Detecting a Central Volume Deficit in Spontaneous Breathing Healthy Volunteers by Systolic Blood Pressure Variation
Brief Title: Detecting a Volume Deficit During Spontaneous Breathing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Michael Dahl, MD, Aalborg University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: H-4-2010-110-SPV
Record Dates: First submitted 2015-09-10; First posted 2015-09-15 (Estimated); Last update posted 2015-09-15 (Estimated); Status verified 2015-09

CONDITIONS: Hypovolemia
Keywords: Central volume deficit; Head-up tilt; Systolic pressure variation
MeSH Terms: conditions — Hypovolemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Respiratory resistor — The volunteers are breathing through the four respiratory resistors (inspiratory, expiratory, combined in- and expiratory and no resistor) in order to increase the intrathoracic pressure svings

SUMMARY:
13 healthy volunteers (4 females) were tilted 45° head-up while breathing through a facemask fitted with an inspiratory and expiratory resistor. A brachial arterial catheter was used to measure blood pressure and thus systolic pressure variation and pulse contour analysis determined stroke volume and thereby cardiac output in order to detect a central volume deficit.

DETAILED DESCRIPTION:
Thirteen healthy volunteers (4 women) at an age of 25 years (range 18-36) were recruited through www.forsøgsperson.dk.

The volunteers were placed on a tilt table and provided with a facemask with an opening of 30-33 mm. A Hook ring was fitted with an inspiratory resistor, an expiratory resistor, a combination of the two resistors, or with no resistance and each resistor provides a 7.5 cmH2O threshold resistance. Each resistor was applied for two minutes with variables obtained in the last minute. The table was then tilted 45° head-up to accumulating blood in the legs and therefore a reduction in the central blood volume. Conversely, 20° head-down tilt was used to expand the central blood volume. For each volunteer measurements with the four respiratory interventions was randomized, whereas the tilt table position was in fixed order: supine, head-up tilt, and head-down tilt.

Three-lead ECG recorded heart rate. A 20 G arterial catheter was placed in the brachial artery of the non-dominant arm and connected to a transducer for reading of blood pressure and stroke volume variation (Vigileo-Flotrac™, version 1.07, Edwards Lifesciences, Nyon, Switzerland). Also SV and CO variation and the arterial pressure curve were recorded for subsequent determination of arterial pressure variations. Additionally, a catheter was placed via a brachial vein to the superior caval vein for recording of central venous pressure and SvO2. While the subjects were breathing spontaneously, the respiratory rate was measured by capnography and peripheral oxygen saturation by fingerprobe.

Variation in the arterial pulse pressure (PPV) was 100 x ((PPmax - PPmin) / ((PPmax + PPmin)/2)), where PPmax and PPmin is the maximal and minimal difference between systolic and diastolic pressure during the respiratory cycle, respectively. By the same formula systolic pressure variation (SPV) was calculated.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers

Exclusion Criteria:

* pregnancy
* lactating
* any regular or acute use of medicine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2011-08; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Systolic pressure variation (SPV) | Two minutes
  Relative difference between systolic blood pressure during inspiration and expiration. Meassured in percent.

REFERENCES:
- [Derived] Dahl M, Hayes C, Steen Rasmussen B, Larsson A, Secher NH. Can a central blood volume deficit be detected by systolic pressure variation during spontaneous breathing? BMC Anesthesiol. 2016 Aug 11;16(1):58. doi: 10.1186/s12871-016-0224-z. PMID 27515038